CLINICAL TRIAL: NCT02475044
Title: Mild Traumatic Brain Injuries in Children: Predicting Behavioral and Emotional Deficits
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rabin Medical Center (Other)
Collaborators: The Israeli insurance companies organization (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 0439-14
Record Dates: First submitted 2015-06-08; First posted 2015-06-18 (Estimated); Last update posted 2016-10-11 (Estimated); Status verified 2016-10

CONDITIONS: Post-Concussion Syndrome
Keywords: post-concussion; Cognitive-Behavioral Theray; parenting
MeSH Terms: conditions — Post-Concussion Syndrome | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment as usual (TAU) (No Intervention): Participants recive Psycho-education and neuro-psycological diagnosis.
- Cognitive-Behavioral Therapy (CBT) (Experimental): Participants recive 16 sessions of CBT in addition to arm TAU treatment.
  Interventions: Behavioral: Cognitive-Behavioral Therapy

INTERVENTIONS:
Behavioral: Cognitive-Behavioral Therapy — 16 Sessions of CBT.
  Other Names: CBT
  Arms: Cognitive-Behavioral Therapy (CBT)

SUMMARY:
The purpose of this study is to investigate the role of psychosocial factors in creating Persistent Post-concussive symptoms (PPCS). The researchers investigate three hypotheses: (a) Do pre-injury psycho-environmental deficits predict a higher level of PPCS? (b) Do socio-demographic and personal pre-injury deficits relate to (1) a more negative attribution for the child injury by their parents and (2) embracing of a more permissive and authoritarian parenting; and do these factors mediate the symptoms' preservation? (c) Does Cognitive-Behavioral Therapy (CBT) benefit to reducing PPCS emotional and behavioral symptoms?

DETAILED DESCRIPTION:
200 children and adolescents with post concussion will be followed for 9 months, since the time of the head injury. Post concussive symptoms, along emotional distress and neurocognitive deficits will be examined at 2 weeks, 4 months and 9 months since the injury, using self report questionnaires, psychological evaluation and neuropsychological tests. Participants who demonstrates PPCS 4 months after the injury will be assigned either to the Cognitive Behavioral Treatmet group (CBT) or to the Treatment as Ususal group(TAU). The change in symptoms severity (PCS, emotional distress and neurocognitive deficits) will be compared between the two study groups in order to assess treatment efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Head trauma.
* Post-concussive symptoms diagnosis according to DSMIV.

Exclusion Criteria:

* mental retardation.
* drug abuse.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 200 (Estimated)
Dates: Start 2015-06; Primary Completion 2018-06 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in the Post Concussion Symptoms Scale at treatment completion. | Approximately 9 months since injury.
  PCI-I (Mittenberg, Miller & Luis, 1997)

SECONDARY OUTCOMES:
Change from Baseline in The State-Trait Anxiety Inventory for Children at Treatment Completion | Approximately 9 months since injury.
  The State-Trait Anxiety Inventory for Children, Spielberger et al.
Change from Baseline in the Childrens Depression Inventory at Treatment Completion | Approximately 9 months since injury.
  Childrens Depression Inventory, Kovacs, 1992
Change from Baseline in The Child PTSD Symptoms Scale at Treatment Completion | Approximately 9 months since injury.
  The Child PTSD Symptoms Scale (Foa et al., 2001)
Change from Baseline in Neuropsychological Functioning at Treatment Subjects will take paper and pencil and computer tests to evaluate memory, learning, attention and concentration, vocabulary and naming. | Approximately 9 months since injury.
  The neuropsychological testing battery includes: Raven's Progressive Matrices, BRIEF, WISC-III-Hebrew Version (Digit Span), CMS (Spatial Span), D-KEFS (Design Fluency, Sorting Test, Trails Making Test), CPT, Stroop,TOMM Effort validity test, The Connors Rating Scale- Revised Long version

CONTACTS AND LOCATIONS:
Overall Officials: Orit Krispin, PhD, Principal Investigator — Schneider Childrens' Medical Center of Israel
Locations (1):
- Schneider Childrens' Medical Center of Israel, Petah Tikva, Israel

IPD SHARING:
Plan to Share IPD: No